CLINICAL TRIAL: NCT03396315
Title: Bisphosphonates for Prevention of Post-Denosumab Bone Loss in Premenopausal Women With Idiopathic Osteoporosis
Brief Title: Bisphosphonates for Prevention of Post-Denosumab Bone Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Elizabeth Shane, Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAR5220
Record Dates: First submitted 2018-01-05; First posted 2018-01-10 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: IOP; Osteoporosis
Keywords: premenopausal women
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: open-label study in which they would choose whether to take oral alendronate 70 mg weekly for 12 months or a single intravenous dose of zoledronic acid 5 mg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- alendronate (Active Comparator): Subjects will receive oral alendronate
  Interventions: Drug: Alendronate
- zoledronic acid (Active Comparator): Subjects will receive zoledronic acid
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Alendronate — oral alendronate 70 mg weekly for 12 months will be given for the prevention of osteoporosis
  Other Names: fosamax
  Arms: alendronate
Drug: Zoledronic Acid — single intravenous dose of zoledronic acid 5 mg will be given for the prevention of osteoporosis
  Other Names: Reclast
  Arms: zoledronic acid

SUMMARY:
The primary goal of the study is to assess the extent to which bisphosphonate therapy will prevent decreases in bone mass that may occur after cessation of denosumab in premenopausal women with idiopathic osteoporosis (IOP) enrolled in AAAN0161 (FD05114) "Denosumab for the prevention of post-teriparatide bone loss in premenopausal women with idiopathic osteoporosis".

In addition, the investigator will observe participants for a second year off bisphosphonate therapy to assess duration of response.

The hypothesis is that bisphosphonate therapy with alendronate or zoledronic acid, initiated after recovery of bone remodeling activity, will prevent significant bone loss after discontinuing denosumab.

DETAILED DESCRIPTION:
Osteoporosis in premenopausal women with normal menstrual function and no specific cause is termed idiopathic osteoporosis (IOP). IOP is a rare disease with an estimated prevalence of <200,000 affected premenopausal women in the United States.

Women with IOP completing at least one year and up to three years of denosumab (Protocol AAAN0161) will be offered participation in this open-label study in which they would choose whether to take oral alendronate 70 mg weekly for 12 months or a single intravenous dose of zoledronic acid 5 mg. Subjects and study personnel will be blinded to BMD outcomes until 12 months.

Discontinuation of denosumab is followed by substantial increases in bone turnover markers to well above baseline, bone resorption reaching twice baseline levels for about 6 months. Over the first 12 months off therapy, all the bone density gained on treatment is lost. Studies done at the institution has demonstrated the occurrence of multiple vertebral fractures in some patients who have stopped denosumab. Based upon these new fracture data, the Prolia label is currently recommending that consideration should be given to transition to another antiresorptive drug in patients stopping denosumab. The main goals of this extension study are to determine rates of bone loss and incidence of radiographic vertebral fractures during one year of bisphosphonate therapy (oral alendronate or intravenous zoledronic acid) initiated after completing denosumab.

ELIGIBILITY:
Inclusion Criteria:

* All women completing at least 12 months of Forteo treatment and at least 12 months of denosumab under previous research studies who remain without a diagnosis of an excluded medical condition and medication exposures as detailed below, will be offered enrollment into this study.

Exclusion Criteria:

* Known intolerance to calcium supplements
* Contraindications to bisphosphonate treatment:

  1. Hypocalcemia
  2. Pregnancy
  3. Known hypersensitivity to bisphosphonates
* History of osteomalacia
* History of osteonecrosis of the jaw
* History of dental extraction or other invasive dental surgery within the prior 4 weeks
* Invasive dental work planned in the next 12 months
* Any condition or illness (acute, chronic, or history), which in the opinion of the Investigator might interfere with the evaluation of efficacy and safety during the study or may otherwise compromise the safety of the subject
* Self-reported or known alcohol or drug abuse within the previous 12 months
* Current or recent (within 1 year of enrollment) inflammatory bowel disease or malabsorption
* Abnormal laboratory tests performed during Visit 1

  1. Renal insufficiency or liver disease: estimated glomerular filtration rate (eGFR) < 35 ml/min, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >50% above upper limit of normal
  2. Hypercalcemia, hypocalcemia
  3. Vitamin D deficiency: 25-Hydroxyvitamin D (25-OHD) < 30 ng/mL
* Subjects must be willing to participate voluntarily. Specifically excluded are the following: 1) women less than 20 (or 35 in the case of those who wish to participate because they have low BMD); 2) protected individuals (institutionalized); 3) prisoners; 4) any other prospective participant who, for any reason, might not be able to give voluntary informed consent.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shane, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Creighton University, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cohen A, Recker RR, Lappe J, Dempster DW, Cremers S, McMahon DJ, Stein EM, Fleischer J, Rosen CJ, Rogers H, Staron RB, Lemaster J, Shane E. Premenopausal women with idiopathic low-trauma fractures and/or low bone mineral density. Osteoporos Int. 2012 Jan;23(1):171-82. doi: 10.1007/s00198-011-1560-y. Epub 2011 Mar 2. PMID 21365462
- [Background] Cohen A, Dempster DW, Recker RR, Stein EM, Lappe JM, Zhou H, Wirth AJ, van Lenthe GH, Kohler T, Zwahlen A, Muller R, Rosen CJ, Cremers S, Nickolas TL, McMahon DJ, Rogers H, Staron RB, LeMaster J, Shane E. Abnormal bone microarchitecture and evidence of osteoblast dysfunction in premenopausal women with idiopathic osteoporosis. J Clin Endocrinol Metab. 2011 Oct;96(10):3095-105. doi: 10.1210/jc.2011-1387. Epub 2011 Aug 10. PMID 21832117
- [Background] Cohen A, Lang TF, McMahon DJ, Liu XS, Guo XE, Zhang C, Stein EM, Dempster DW, Young P, Saeed I, Lappe JM, Recker RR, Shane E. Central QCT reveals lower volumetric BMD and stiffness in premenopausal women with idiopathic osteoporosis, regardless of fracture history. J Clin Endocrinol Metab. 2012 Nov;97(11):4244-52. doi: 10.1210/jc.2012-2099. Epub 2012 Sep 7. PMID 22962425
- [Background] Cohen A, Liu XS, Stein EM, McMahon DJ, Rogers HF, Lemaster J, Recker RR, Lappe JM, Guo XE, Shane E. Bone microarchitecture and stiffness in premenopausal women with idiopathic osteoporosis. J Clin Endocrinol Metab. 2009 Nov;94(11):4351-60. doi: 10.1210/jc.2009-0996. Epub 2009 Oct 16. PMID 19837923
- [Background] Cohen A, Stein EM, Recker RR, Lappe JM, Dempster DW, Zhou H, Cremers S, McMahon DJ, Nickolas TL, Muller R, Zwahlen A, Young P, Stubby J, Shane E. Teriparatide for idiopathic osteoporosis in premenopausal women: a pilot study. J Clin Endocrinol Metab. 2013 May;98(5):1971-81. doi: 10.1210/jc.2013-1172. Epub 2013 Mar 29. PMID 23543660
- [Background] Nishiyama K, Wang J, Young P, et al. Teriparatide Is Associated with Improved Microarchitecture and Estimated Bone Strength in Premenopausal Women with Idiopathic Osteoporosis: An HR-pQCT Study. American Society for Bone and Mineral Research Annual Meeting; 2013; Baltimore, MD: American Society for Bone and Mineral Research
- [Background] Cosman F, Nieves J, Woelfert L, Formica C, Gordon S, Shen V, Lindsay R. Parathyroid hormone added to established hormone therapy: effects on vertebral fracture and maintenance of bone mass after parathyroid hormone withdrawal. J Bone Miner Res. 2001 May;16(5):925-31. doi: 10.1359/jbmr.2001.16.5.925. PMID 11341338
- [Background] Lane NE, Sanchez S, Modin GW, Genant HK, Pierini E, Arnaud CD. Parathyroid hormone treatment can reverse corticosteroid-induced osteoporosis. Results of a randomized controlled clinical trial. J Clin Invest. 1998 Oct 15;102(8):1627-33. doi: 10.1172/JCI3914. PMID 9788977
- [Background] Lane NE, Sanchez S, Modin GW, Genant HK, Pierini E, Arnaud CD. Bone mass continues to increase at the hip after parathyroid hormone treatment is discontinued in glucocorticoid-induced osteoporosis: results of a randomized controlled clinical trial. J Bone Miner Res. 2000 May;15(5):944-51. doi: 10.1359/jbmr.2000.15.5.944. PMID 10804025
- [Background] Finkelstein JS, Arnold AL. Increases in bone mineral density after discontinuation of daily human parathyroid hormone and gonadotropin-releasing hormone analog administration in women with endometriosis. J Clin Endocrinol Metab. 1999 Apr;84(4):1214-9. doi: 10.1210/jcem.84.4.5643. PMID 10199756
- [Background] Cohen A, Kamanda-Kosseh M, Recker RR, Lappe JM, Dempster DW, Zhou H, Cremers S, Bucovsky M, Stubby J, Shane E. Bone Density After Teriparatide Discontinuation in Premenopausal Idiopathic Osteoporosis. J Clin Endocrinol Metab. 2015 Nov;100(11):4208-14. doi: 10.1210/jc.2015-2829. Epub 2015 Sep 10. PMID 26358172
- [Background] Bone HG, Bolognese MA, Yuen CK, Kendler DL, Miller PD, Yang YC, Grazette L, San Martin J, Gallagher JC. Effects of denosumab treatment and discontinuation on bone mineral density and bone turnover markers in postmenopausal women with low bone mass. J Clin Endocrinol Metab. 2011 Apr;96(4):972-80. doi: 10.1210/jc.2010-1502. Epub 2011 Feb 2. PMID 21289258
- [Background] Miller PD, Bolognese MA, Lewiecki EM, McClung MR, Ding B, Austin M, Liu Y, San Martin J. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone. 2008 Aug;43(2):222-229. doi: 10.1016/j.bone.2008.04.007. Epub 2008 Apr 26. PMID 18539106
- [Background] Anastasilakis AD, Makras P. Multiple clinical vertebral fractures following denosumab discontinuation. Osteoporos Int. 2016 May;27(5):1929-30. doi: 10.1007/s00198-015-3459-5. Epub 2015 Dec 22. No abstract available. PMID 26694593
- [Background] Anastasilakis AD, Polyzos SA, Makras P, Aubry-Rozier B, Kaouri S, Lamy O. Clinical Features of 24 Patients With Rebound-Associated Vertebral Fractures After Denosumab Discontinuation: Systematic Review and Additional Cases. J Bone Miner Res. 2017 Jun;32(6):1291-1296. doi: 10.1002/jbmr.3110. Epub 2017 Mar 13. PMID 28240371
- [Background] Anastasilakis AD, Yavropoulou MP, Makras P. Bisphosphonates or denosumab discontinuation and risk of fractures. Maturitas. 2017 Aug;102:75. doi: 10.1016/j.maturitas.2017.04.016. Epub 2017 Apr 27. No abstract available. PMID 28495014
- [Background] Anastasilakis AD, Yavropoulou MP, Makras P, Sakellariou GT, Papadopoulou F, Gerou S, Papapoulos SE. Increased osteoclastogenesis in patients with vertebral fractures following discontinuation of denosumab treatment. Eur J Endocrinol. 2017 Jun;176(6):677-683. doi: 10.1530/EJE-16-1027. Epub 2017 Mar 10. PMID 28283537
- [Background] Aubry-Rozier B, Gonzalez-Rodriguez E, Stoll D, Lamy O. Severe spontaneous vertebral fractures after denosumab discontinuation: three case reports. Osteoporos Int. 2016 May;27(5):1923-5. doi: 10.1007/s00198-015-3380-y. Epub 2015 Oct 28. PMID 26510845
- [Background] Lamy O, Gonzalez-Rodriguez E, Stoll D, Hans D, Aubry-Rozier B. Severe Rebound-Associated Vertebral Fractures After Denosumab Discontinuation: 9 Clinical Cases Report. J Clin Endocrinol Metab. 2017 Feb 1;102(2):354-358. doi: 10.1210/jc.2016-3170. PMID 27732330
- [Background] Popp AW, Zysset PK, Lippuner K. Rebound-associated vertebral fractures after discontinuation of denosumab-from clinic and biomechanics. Osteoporos Int. 2016 May;27(5):1917-21. doi: 10.1007/s00198-015-3458-6. Epub 2015 Dec 22. PMID 26694598
- [Background] Freemantle N, Satram-Hoang S, Tang ET, Kaur P, Macarios D, Siddhanti S, Borenstein J, Kendler DL; DAPS Investigators. Final results of the DAPS (Denosumab Adherence Preference Satisfaction) study: a 24-month, randomized, crossover comparison with alendronate in postmenopausal women. Osteoporos Int. 2012 Jan;23(1):317-26. doi: 10.1007/s00198-011-1780-1. Epub 2011 Sep 17. PMID 21927922
- [Background] Reid IR, Horne AM, Mihov B, Gamble GD. Bone Loss After Denosumab: Only Partial Protection with Zoledronate. Calcif Tissue Int. 2017 Oct;101(4):371-374. doi: 10.1007/s00223-017-0288-x. Epub 2017 May 13. PMID 28500448
- [Derived] Cohen A, Kamanda-Kosseh M, Rawal R, Agarwal S, Barry J, Shiau S, Colon I, Bucovsky M, Lappe JM, Shane E. Bone density and remodeling after discontinuation of sequential therapy for premenopausal idiopathic osteoporosis. Osteoporos Int. 2025 Dec 14. doi: 10.1007/s00198-025-07755-z. Online ahead of print. PMID 41392041
- See also: Department of Endocrinology at Columbia University — http://columbiamedicine.org/divisions/Endo/index.shtml

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alendronate | Zoledronic Acid
Started | 18 | 6
Completed | 18 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alendronate | Zoledronic Acid | Total
Number analyzed (Participants) | 18 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 6 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (8.6) | 34.7 (6.3) | 37.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 6 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 6 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Difference in BMD at the Lumbar Spine (L1-4) Within Group
Description: Within-group difference (percent change) in BMD at the lumbar spine (L1-4) will be measured by Dual-energy X-ray absorptiometry (DXA) and calculated.
Time Frame: Baseline, 12 month
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Alendronate | Zoledronic Acid
Number analyzed (Participants) | 18 | 6
percentage of change | -1.1 (4.8) | -2.4 (1.0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Alendronate | Zoledronic Acid
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6
Other Adverse Events (participants affected / at risk) | 12/18 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alendronate (N=18) | Zoledronic Acid (N=6)
Acute phase reaction (Immune system disorders) | 0 (0) | 5 (5)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Covid (Immune system disorders) | 0 (0) | 1 (1)
Numbness (Nervous system disorders) | 1 (1) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hot flashes (Endocrine disorders) | 3 (3) | 0 (0)
Acid regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT03396315/Prot_SAP_000.pdf